CLINICAL TRIAL: NCT07028515
Title: Effects of Self-controlled Practice on Motor Learning and Motivation in People With Parkinson's Disease
Brief Title: Self-controlled Practice on Motor Learning and Motivation in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202503040RINA
Record Dates: First submitted 2025-06-08; First posted 2025-06-19 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; motor learning; motivation; self-controlled practice
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PD self-controlled group: PD participants in the choice condition
- PD yoked group: PD participants in the no-choice condition
- HC self-controlled group: Healthy controls in the choice condition
- HC yoked group: Healthy controls in the no-choice condition

SUMMARY:
People with Parkinson's disease have been known to have low motivation and motor learning impairment, which might limit the effectiveness of neurorehabilitation, exacerbate motor performance and quality of life, and increase the burden on caregivers. Therefore, enhancing motor learning ability and motivation is crucial for people with PD. According to the OPTIMAL theory, practice under self-controlled conditions has been shown to improve motivation and learning in healthy individuals. However, few studies have explored the effects of self-controlled practice on motor learning and motivation in people with PD and examined the underlying neurophysiological mechanisms. This study aims to investigate the effects of self-controlled practice on motor learning and motivation in people with PD, as well as the associated neurophysiological changes.

People with PD and age-matched healthy controls without neurological disorders will be recruited. Participants will be pair-matched based on age, gender, and disease severity, and then assigned to either the self-controlled group or the yoked group. The participants will be required to visit the lab for a total of three times in one week: on Day 1 for baseline assessments, neurophysiological evaluation using transcranial magnetic stimulation (TMS), practice of the trajectory matching task, motivation evaluation, and exercise education; on Day 2 for additional trajectory matching task practice, motivation evaluation, immediate retention test of the task, neurophysiological evaluation using TMS, and exercise education; and on Day 7 for delayed retention and transfer tests and final TMS assessment. On Days 1 and 2, all participants will practice the trajectory matching task. At the beginning of each trial, a target trajectory will be shown, and participants will be asked to replicate it using a joystick. Feedback will be provided after each trial to indicate accuracy. The self-controlled group will be allowed to choose the story contents they prefer when practicing the task, and the exercise they would like to learn after the task. In contrast, yoked participants will receive the same story and exercise education as their matched counterparts in the self-controlled group.

This study will help clarify the effects of self-controlled practice on motor learning and motivation in people with PD, offering a new perspective for clinical interventions and emphasizing the importance of patients actively participating in treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* age above 20-year-old
* able to follow instructions and the rules of the motor task
* do not have surgery or injury in their upper extremities in the past 6 months

Exclusion Criteria:

* neurological disorders other than PD
* symptoms of severe tremor in upper extremities
* symptoms of anxiety and depression
* deep brain stimulator or pacemaker implanted in the body
* history of seizure or epilepsy
* unstable medical conditions
* migraines or tinnitus uncontrolled by medication
* pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with PD are idiopathic PD diagnosed by a neurologist. Healthy controls are without any neurological disorders.
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Root mean square error (RMSE) | Day 1 (practice phase), day 2 (practice phase and immediate retention), and day 7 (delayed retention and transfer)
  The accuracy of the overall performance of the target waveform trajectory. The RMSE is the mean difference between the target waveform trajectory and the participant's performed waveform trajectory calculated over their actual movement time. Smaller RMSE value indicates better task performance. With a total of 144 trials practiced during the practice phase on D1 and D2, the RMSE will be averaged every 12 trials as a block for later data analysis and presentation, resulting in a total of 12 practice blocks (B1 to B12), 2 retention test blocks (imme-ret and delay-ret) and 1 transfer test block (xfer).

SECONDARY OUTCOMES:
Error estimation (EE) test | Day 2 (immediate retention) and day 7 (delayed retention and transfer)
  The participants will be required to verbally estimate their RMSE after each trial for retention and transfer test trials. The equation for calculating EE is √(CE^2+ VE^2 ), while constant error (CE) captures estimation bias (estimated-actual) and variable error (VE) is the standard deviation of these errors. A lower EE value indicates that the participants are more precise in estimating their performance and suggests better cognitive processing.
Motivation evaluation | Day 1 and 2
  Motivation evaluation will be conducted after the practice phase during day 1 and day 2, and will be assessed with a self-reported motivational questionnaire consisting of perceived competence, task interest/enjoyment, and autonomy. This motivation questionnaire is composed of a total of 14 items scored on a 7-point Likert scale. Score ranges from 14 to 98, with a higher score indicating better perceived competence, task interest/enjoyment, and autonomy.
Transcranial magnetic stimulation (TMS) assessment | Day 1, 2, and 7
  TMS is a non-invasive neurophysiological assessment tool used to evaluate changes in corticomotor excitability associated with self-controlled practice in motor learning. Assessments will be conducted using the Magstim® BiStim² (The Magstim Company Ltd., Whitland, UK) device with a figure-of-eight coil. TMS outcomes of interest will include resting and active motor-evoked potential (MEP), cortical silent period (CSP), short-interval intracortical inhibition (SICI), and intracortical facilitation (ICF).
Movement Disorder Society Unified Parkinson's Disease Rating Scale | Day 1
  It consists of 4 parts, including non-motor aspects of experiences of daily living, motor aspects of experiences of daily living, motor examination, and motor complications. Total score ranges from 0 to 200, with a higher score indicating greater disease severity.
Apathy Evaluation Scale | Day 1
  The Chinese version of the self-rated Apathy Evaluation Scale (AES) will be used to measure apathy. Each item scores on a 4-point Likert scale, and the score ranges from 18 to 72, with a higher score indicating greater apathy.
short-form Lille Apathy Rating Scale | Day 1
  The clinician-rated short-form Lille Apathy Rating Scale (short-form LARS) will be used to measure apathy. The scale is scored with a 5-point Likert scale in the first 3 items and a binary (yes/no) scale with an additional "not available (NA)" condition for non-classifiable or non-applicable answers or items. The total score ranges between -15 and 15, with a higher score indicating greater severity in apathy.
Montreal Cognitive Assessment (MoCA) | Day 1
  Cognitive function of the participants will be assessed through Montreal Cognitive Assessment (MoCA), which is a widely used screening tool for detecting cognitive impairment. The MoCA consists of memory, attention, language, abstraction, orientation to time and place, visuospatial abilities, and executive functions. The total score ranges from 0 to 30, with a higher score indicating better cognitive function.
Hospital Anxiety and Depression Scale (HADS) | Day 1
  Hospital Anxiety and Depression Scale (HADS) will be conducted for evaluating the symptoms of anxiety and depression. The HADS consists of 14 items, which 7 items are categorized into anxiety (HADS-A) and 7 items into depression (HADS-D). Each item will be scored on a 4-point Likert scale with a total score ranging from 0 to 21, and a higher score indicates greater symptoms of anxiety and depression. The cutoff score for identifying symptoms of anxiety and depression in the PD population has been established as ≥ 11 points in the anxiety or depression subscales, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Graduate Institute of Physical Therapy, Principal Investigator — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, Taipei, Zhongzheng Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewthwaite R, Chiviacowsky S, Drews R, Wulf G. Choose to move: The motivational impact of autonomy support on motor learning. Psychon Bull Rev. 2015 Oct;22(5):1383-8. doi: 10.3758/s13423-015-0814-7. PMID 25732095
- [Background] Wulf G, Lewthwaite R. Optimizing performance through intrinsic motivation and attention for learning: The OPTIMAL theory of motor learning. Psychon Bull Rev. 2016 Oct;23(5):1382-1414. doi: 10.3758/s13423-015-0999-9. PMID 26833314
- [Background] Chiviacowsky S, Wulf G, Lewthwaite R, Campos T. Motor learning benefits of self-controlled practice in persons with Parkinson's disease. Gait Posture. 2012 Apr;35(4):601-5. doi: 10.1016/j.gaitpost.2011.12.003. Epub 2011 Dec 30. PMID 22209649